CLINICAL TRIAL: NCT06217510
Title: Pilot Project on the Automatic Design and 3D Printing of Adolescent Idiopathic Scoliosis Braces (Phase 1)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: Modulate Technologies (Unknown)
Responsible Party: Principal Investigator, Hubert Labelle, MD, Orthopeadic Surgeon, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-21-2024-6669
Record Dates: First submitted 2024-01-08; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; 3D printing; Finite Element Analysis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: Pilot study with a single group of 15 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Brace (Experimental): A 3D printed brace designed automatically from a digital twin of the participant.
  Interventions: Device: Test Brace

INTERVENTIONS:
Device: Test Brace — Participants will be fitted with the Test Brace and will wear the brace for 30 minutes.

SUMMARY:
The goal of this pilot clinical trial is to validate a 3D printed brace designed automatically for patients with Adolescent Idiopathic Scoliosis. The main question it aims to answer is: which parameters leads to a efficient and comfortable brace.

Participants will try the brace for a period of 30 minutes, measurement and feedback will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of Adolescent Idiopathic Scoliosis
* Risser 0-2
* Cobb Angle between 20 and 40 degrees
* Prescription for a brace
* Able to understand French or English

Exclusion Criteria:

* Grade II or higher Spondylolisthesis
* Neuromuscular disease
* Past spinal surgery

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Participant Questionnaire | 30 minutes
  Questionnaire given to the participant after the testing period. Data about the experience, impressions about the brace and the comfort will be recorded.
Orthotist Adjustment Questionnaire | 30 minutes
  Questionnaire given to the orthotist after the testing period. Data about the number of adjustment and his experience working with the brace will be recorded.

IPD SHARING:
Plan to Share IPD: No